CLINICAL TRIAL: NCT07278934
Title: Testing the Impact of Family-Based Intervention to Improve Developmental and Health Outcomes for Female Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: University of Ghana (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD116780 (NIH)
Record Dates: First submitted 2025-12-06; First posted 2025-12-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Unaccompanied Migration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolstered care (No Intervention): Female adolescents in the bolstered care will receive services/education as usual in their respective schools. The usual care will be bolstered by providing school supplies (e.g., textbooks, notebooks)
- ANZANSI Family Program (Experimental): In addition to bolstered care, participants in this arm will receive the ANZANSI intervention comprised of family economic empowerment (FEE) intervention and multiple family group (MFG) intervention. FEE includes: 1) Financial Literacy Training; 2) Child Development Account (CDA); and 3) Family income-generating/microenterprise promotion component
  Interventions: Behavioral: ANZANSI Family Program

INTERVENTIONS:
Behavioral: ANZANSI Family Program — Family Economic Empowerment: 1) Financial literacy training: Four 1-2 hour workshop sessions focused on financial literacy will be delivered. 2) CDA. Each participant receives a CDA, a matched savings account. Participants' family members, relatives, or friends are allowed and encouraged to contribute towards the CDA. The account is then matched with money from the project. The match cap is an equivalent of US$10 per month; 3) The family income-generating activity (IGA): Participants are trained on IGAs and expected to use part of their matched savings to start an IGA.
  Multiple Family Groups. The manualized 16-session intervention is organized around 4Rs (Rules, Responsibility, Relationships, and Respectful Communication) and 2Ss (Stress and Social Support). Children and caregivers complete activities together or split to reconvene later for discussing as a larger group. Each group involves 7 to 10 families, with at least two generations of a family present in each session.
  Arms: ANZANSI Family Program

SUMMARY:
This study seeks to address the urgent need for theoretically and empirically informed interventions that would address the increasing numbers of unaccompanied minors migrating from rural to urban centers in developing countries for better economic opportunities. This process often results in hazardous child labor defined as work that is mentally, physically, socially or morally dangerous and harmful; interfering with schooling and health and mental health functioning, and leading to several other disproportionate risks. Unaccompanied migrant child laborers' vulnerability is further intensified by the lack of parental protection and community belonging in the host urban center. The International Labor Organization (ILO) estimates that 9.6% of children (ages 5 to 17) across the globe are child laborers and draws attention to migrant child laborers as an underreported and highly vulnerable group, a significant portion of which are female with no education. Poverty has been identified as the main driver of child labor, with family context also being a critical contributing factor. Sub-Saharan Africa (SSA) has the highest rates of child labor (24%), with Ghana -the focus of this study- registering one of the highest child labor prevalence at 22%, including unaccompanied child migrant laborers. In Ghana, unaccompanied adolescent girls migrate from the Northern region to urban centers in the south to work in the informal economy. Load carrying is the most common type of labor for this population and exposes migrant girls to multiple developmental and health risks. Building on the recently concluded R21 study (with 97 adolescent girls aged 11 to 14 years and their caregivers) that showed high feasibility and acceptability, and promising preliminary impact of the ANZANSI (resilience in Dagbani -local language) combination intervention in the same region, we propose to test its effectiveness in a larger two-arm cluster randomized clinical trial among 960 adolescent girls (age 11 to 14 years) at risk of school dropout nested within 32 public junior high schools in the Northern region of Ghana and their caregivers. The schools will be randomly assigned to one of two study conditions: 1) ANZANSI (FEE+MFG) and 2) bolstered usual care. The intervention will be delivered for 12 months, with assessments conducted at baseline and at 12-, 24-, and 36-month follow-ups post-intervention initiation. The study specific aims are: Aim 1: Examine the short- and medium-term impacts of ANZANSI intervention on the incidence of unaccompanied migration for child labor (primary outcome), and academic progress and psychosocial outcomes (secondary); Aim 2: Examine the impact of the ANZANSI intervention on potential mechanisms of change at the individual, family, and community levels; Aim 3: Evaluate the cost and cost-effectiveness of each intervention condition; and Aim 4: Qualitatively examine participants, facilitators, and school leadership's experiences with the intervention.

ELIGIBILITY:
Inclusion Criteria:

Adolescent girls' inclusion criteria are:

* Enrolled in school and living within a family (defined broadly -not necessarily biological parents)
* Ages 11 to 14
* Skipping school in the past academic term (with at least 10% of unexcused absences).
* Capable of giving assent

The caregiver inclusion criteria

* Age 18 or older
* Self-identified as primary caregiver of the adolescent girl
* Capable of providing informed consent.

Exclusion Criteria:

- Participants that do not meet the criteria or exhibit a lack of understanding of the study procedures and hence not able to provide informed consent will be excluded.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1920 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2030-08-15 (Estimated); Study Completion 2030-08-15 (Estimated)

PRIMARY OUTCOMES:
Unaccompanied migration | 12 months, 24 months, 36 months
  Change in the incidence of unaccompanied migration will be measured by a two-item scale (yes/no) and school records

SECONDARY OUTCOMES:
Self-concept | baseline, 12 months, 24 months, 36 months
  Change in self-concept will be measured by the Tennessee Self-Concept Scale Short Form. The 20-item short version of the original 100-item TSCS scale assesses adolescents' perception of self-identity and self-satisfaction. The items are rated on a 5-point Likert scale ranging from 1 = always false to 5 = always true. The theoretical range for the TSCS was 20-100, with higher scores representing a more positive self-concept.
self-esteem | baseline, 12 months, 24 months, 36 months
  Change in self-esteem will be measured using Rosenberg's self-esteem scale (RSES). The scale comprises 10 statements about general feelings of self-worth or self-acceptance rated on a 4-point Likert scale response option (strongly agree to strongly disagree, with 4 = strongly agree, 3 = agree, 2 = disagree, 1 = strongly disagree). The items were scored on a theoretical range of 10-40 and summed, with higher scores representing higher self-esteem.
life satisfaction | baseline, 12 months, 24 months, 36 months
  Change in life satisfaction will be measured using the multi-dimensional student life satisfaction scale (MSLSS). The scale includes 40 items assessing life satisfaction on 5 specific aspects while maintaining an overall life satisfaction score. Responses are rated on a 6-point Likert scale with 1 = strongly disagree, 2 = moderately disagree, 3 = slightly disagree, 4 = slightly agree, 5 = moderately agree, and 6 = strongly agree (theoretical range 40-240). Higher values representing higher satisfaction in student life.
school attendance | baseline, 12 months, 24 months, 36 months
  Change in school attendance for the past academic year will be measured using school records.
grade progress | baseline, 12 months, 24 months, 36 months
  Grade progress will be measured using a three-response question (0= enrolled in expected grade, 1=grade repetition, 2=dropout)
attitudes toward school | baseline, 12 months, 24 months, 36 months
  Change in attitudes towards school will be measured by School attitude assessment survey. The range is 20 to 100, with higher scores representing a more positive attitude towards school. Attitudes toward school were assessed using the school attitude assessment survey (SAAS; McCoach, 2002). The survey consists of 20 items rated on a 5-point Likert scale (1 = not at all, 2 = a little bit, 3 = pretty well, 4 = well, and 5 = very well). The scale measures aspects of students' lives that predict their academic achievement, including peer attitudes, attitudes toward school, self-motivation, and self-regulation. Higher values representing higher positive attitudes toward school.
social support | baseline, 12 months, 24 months, 36 months
  change in social support will be measured using the social support behavior scale. The SS-B measure consists of 45 items designed to tap five modes of support: emotional support, socializing, practical assistance, financial assistance, and advice/guidance. The Likert scale is from 1=strongly disagree to 5=strongly agree. The theoretical range is 45-225, with higher scores indicating higher social support.
perceived social support | baseline, 12 months, 24 months, 36 months
  Change in perceived social support will be measured by the Multidimensional Scale of Perceived Social Support. The MSPSS is a self-report measure to assess participants' social support. The 12-item scale had statements such as, "there is a special person who is around when I am in need," rated on a 5-point Likert scale ranging from strongly agree to strongly disagree, with 5=strongly agree, 4=agree, 3=neutral, 2=disagree, 1=strongly disagree. The theoretical range is 12-60, with higher scores indicating greater social support.
family cohesion | baseline, 12 months, 24 months, 36 months
  change in family cohesion will be measured by a 7-item measure adapted from Family environment scale and family assessment measure. The items measure the degree of commitment, help and support family members provide for one another. Participants are asked to rate how often each item occurred in their family using a 5-point scale (with 1 = 'never' and 5 = 'always'). Items include 'Do your family members ask each other for help before asking nonfamily members for help?', and 'Do you listen to what other family members have to say, even when you disagree?' Theoretical range is 7 to 35, with higher scores indicating higher levels of family cohesion.
parenting stress | baseline, 12 months, 24 months, 36 months
  change in parenting stress will be measured by parental stress scale (PSS) developed by Berry and Jones (1995). The 18 item scale is scored with a 5-point likert scale, 1 = Strongly disagree 2 = Disagree 3 = Undecided 4 = Agree 5 = Strongly agree (theoretical range 18-80). Items represent positive (e.g. emotional benefits, personal development) and negative (demands on resources, restrictions) themes of parenthood. Lower scores represent lower levels of parenting stress.
Intention to migrate | baseline, 12 months, 24 months, 36 months
  change in intention to migrate will be measured by one item: How likely do you (the adolescent girl) see yourself migrating? The question uses a likert scale ranging from 1 (very unlikely) to 5 (very likely).
gender norms | baseline, 12 months, 24 months, 36 months
  change in gender norms will be measured by the 10-item scale adapted from the Gender Norm Attitudes Scale (Waszak et al., 2001), which measures participants' understanding of the appropriateness of behaviors as they relate to being female and male. The items in the scale encompass aspects related to educational performance, future expectations for both genders, family support, encouragement, decision-making, and involvement in intimate relationships and behaviors. The scale items featuredbinary responses (Agree = 1 and Disagree = 0; theoretical range 0-10). Higher scores denote more egalitarian gender norms and beliefs.
future orientation | baseline, 12 months, 24 months, 36 months
  change in future orientation will be measured by two items evaluating adolescents' expectations and optimism regarding their educational goals. The first item asks participants, How sure are you that you will achieve your educational plans? with response options ranging from 1 = Not at all sure to 5 = Extremely sure. The second item asks, How hopeful are you that you will achieve your educational plans? with parallel response options ranging from 1 = Not at all hopeful to 5 = Extremely hopeful (theoretical range 2-10). Higher scores indicate a more positive future orientation
confidence in saving | baseline, 12 months, 24 months, 36 months
  change in confidence in saving will be measured by the confidence in saving survey that includes 5 items that assess participant's confidence in saving and saving-related behaviors. The survey uses a 5-point likert scale: 5= extremely confident, 4= very confident, 3= somewhat confident, 2= not very confident, or 1= not confident at all (theoretical range 5-25). Higher scores indicate higher confidence
importance of saving | baseline, 12 months, 24 months, 36 months
  change in importance of saving will be measured by the importance of saving survey that includes 5 items that assess importance of saving for participants. The survey uses a 5-point Likert scale: 5= extremely important, 4= very important, 3= somewhat important, 2= not very important, or 1= not important at all (theoretical range 5-25). Higher scores indicate higher importance of saving for participants.
saving | 12 months, 24 months, 36 months
  change in savings overtime in the intervention group will be measured by monthly bank statements
child-caregiver relationship | baseline, 12 months, 24 months, 36 months
  The perceived child-caregiver relationship scale is adapted from the Family Assessment measure and assess relationships on two dimensions: (1) acceptance and warmth - the extent to which the caregiver perceives as involved in their child's life; and (2) psychological autonomy - the extent to which the caregiver employs a non-coercive, democratic discipline and encourages the child to express individuality within the family. Participants are asked to rate the adults they live with, on each of the 17 items (range: 17-85), on a 5-point scale (1 = 'never' and 5 = 'always'). Sample items include: "Can you count on your parents to help her if she has a problem?" and "Do your parents keep challenging you to do the best in whatever you do?" Higher scores indicatw a more positive child-caregiver relationship.

IPD SHARING:
Plan to Share IPD: Yes
The study team will use the NICHD Data and Specimen Hub (DASH) to deposit the data. DASH is a centralized resource that allows researchers to share and access de-identified data from studies fundedby NICHD.
Supporting Information: SAP
Time Frame: Data will become public after results on the study outcomes are analyzed and published.